CLINICAL TRIAL: NCT03019796
Title: Effects of Exercise Training as a Non-pharmacological Treatment for Metabolic Syndrome and Its Interactions With Subjects Habitual Medications.
Brief Title: Exercise Training Effects on Metabolic Syndrome: Interactions With Medication
Acronym: METSYND
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Castilla-La Mancha (Other)
Collaborators: Ministerio de Economía y Competitividad, Spain (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 0112001154 DEP2014-52930-R
Record Dates: First submitted 2016-12-31; First posted 2017-01-13 (Estimated); Results first posted 2021-05-18 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-05

CONDITIONS: Exercise Therapy; Metabolic Syndrome X; Cardiorespiratory Fitness
MeSH Terms: conditions — Metabolic Syndrome | interventions — Dosage Forms; Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PLACEBO FIRST THEN MEDICATED (Experimental): Subjects first receive the PLACEBO tablet during 72 hours (full withdrawal). After a week of taking again their medication (MEDICATION TRIAL), they will be tested again. This procedure will be repeated before and after 4 months of aerobic training.
  Interventions: Drug: MEDICATION AND EXERCISE TRAINING
- MEDICATED FIRST THEN PLACEBO (Experimental): Subjects first receive their antihypertensive MEDICATION tablet (habitual dose prescribed by their primary care doctors). After a week they will take a PLACEBO tablet for 72 hours and will be tested again. This procedure will be repeated before and after 4 months of aerobic training.
  Interventions: Drug: MEDICATION AND EXERCISE TRAINING

INTERVENTIONS:
Drug: MEDICATION AND EXERCISE TRAINING — PARTICIPANTS WILL BE (IN A RANDOMIZED BLINDED FASHION) WITHDRAWN OF THEIR HYPERTENSIVE MEDICATION (I.E., PLACEBO) IN ONE OCCASION AND TESTED WITH THEIR MEDICATION IN ANOTHER, WITH A WEEK WASHOUT PERIOD.
  THIS TESTING WILL BE REPEATED AFER 4 MONTHS OF EXERCISE TRAINING (48 SESSIONS OF 43 MIN EACH ONE).

SUMMARY:
To analyze the effects of different exercise training modalities (continuous, intervallic, and resistance training) on cardiorespiratory and metabolic fitness of metabolic syndrome patients when this training interacts with their habitual medication.

DETAILED DESCRIPTION:
Objective: The purpose is to study in a group of adults with metabolic syndrome and obesity, the effects of different modalities of exercise training on cardiorespiratory and metabolic fitness. The main objective is to weight the effects of exercise training separately and in conjunction with the subject's habitual pharmacological treatment to identify the best combination of drug and exercise.

Methods and design: Randomized, pretest-posttest control group experimental design. Project developed in a single center with the collaboration of the regional public health system.

Subjects: Will be referred by their primary care physicians to our study unit. Up to 40 subjects all of them with metabolic syndrome will be recruited (at least 20% women).

Measurements:

1. Specifically, the investigators, will study cardiovascular adaptations that increase, i) maximal aerobic capacity measured by VO2max, ii) anaerobic and respiratory compensation point ventilatory thresholds, iii) arterial stiffness, measured by pulse wave velocity (SphygmoCor System), v) central and peripheral blood pressure, and iv) biological markers of endothelial dysfunction using reactive hyperemia with a laser Doppler fluxmeter in central and peripheral blood vessels.
2. The metabolic adaptations under study will include, i) insulin sensitivity by HOMA-IR, ii) fat oxidation by indirect calorimetry

ELIGIBILITY:
Inclusion Criteria:

* Metabolic syndrome patients diagnosed according to the International diabetes federation consensus of 2009 (Alberti, et al., Circulation).
* 18-65 years old

Exclusion Criteria:

Cardiovascular disease or musculo-skeletal that prevents them from being able to perform intense exercise.

* Respiratory failure
* Patient ends
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2020-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Mora-Rodriguez, PhD, Principal Investigator — University of Castilla-La Mancha
Locations (1):
- University of Castilla-La Mancha (Exercise Physiology Lab), Toledo, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Morales-Palomo F, Ramirez-Jimenez M, Ortega JF, Pallares JG, Mora-Rodriguez R. Cardiovascular Drift during Training for Fitness in Patients with Metabolic Syndrome. Med Sci Sports Exerc. 2017 Mar;49(3):518-526. doi: 10.1249/MSS.0000000000001139. PMID 27787335
- [Background] Ortega JF, Morales-Palomo F, Fernandez-Elias V, Hamouti N, Bernardo FJ, Martin-Doimeadios RC, Nelson RK, Horowitz JF, Mora-Rodriguez R. Dietary supplementation with omega-3 fatty acids and oleate enhances exercise training effects in patients with metabolic syndrome. Obesity (Silver Spring). 2016 Aug;24(8):1704-11. doi: 10.1002/oby.21552. Epub 2016 Jun 29. PMID 27356240
- [Background] Mora-Rodriguez R, Ortega JF, Guio de Prada V, Fernandez-Elias VE, Hamouti N, Morales-Palomo F, Martinez-Vizcaino V, Nelson RK. Effects of Simultaneous or Sequential Weight Loss Diet and Aerobic Interval Training on Metabolic Syndrome. Int J Sports Med. 2016 Apr;37(4):274-81. doi: 10.1055/s-0035-1564259. Epub 2015 Dec 14. PMID 26667921
- [Background] Ortega JF, Fernandez-Elias VE, Hamouti N, Pallares JG, Mora-Rodriguez R. Higher Insulin-sensitizing Response after Sprint Interval Compared to Continuous Exercise. Int J Sports Med. 2015 Mar;36(3):e4. doi: 10.1055/s-0035-1548800. Epub 2015 Mar 26. No abstract available. PMID 25811624
- [Background] Martinez-Vizcaino V, Sanchez-Lopez M, Notario-Pacheco B, Salcedo-Aguilar F, Solera-Martinez M, Franquelo-Morales P, Lopez-Martinez S, Garcia-Prieto JC, Arias-Palencia N, Torrijos-Nino C, Mora-Rodriguez R, Rodriguez-Artalejo F. Gender differences on effectiveness of a school-based physical activity intervention for reducing cardiometabolic risk: a cluster randomized trial. Int J Behav Nutr Phys Act. 2014 Dec 10;11:154. doi: 10.1186/s12966-014-0154-4. PMID 25491026
- [Background] Ortega JF, Fernandez-Elias VE, Hamouti N, Pallares JG, Mora-Rodriguez R. Higher insulin-sensitizing response after sprint interval compared to continuous exercise. Int J Sports Med. 2015 Mar;36(3):209-14. doi: 10.1055/s-0034-1389942. Epub 2014 Nov 6. PMID 25376729
- [Background] Ortega JF, Hamouti N, Fernandez-Elias VE, Mora-Rodriguez R. Comparison of glucose tolerance tests to detect the insulin sensitizing effects of a bout of continuous exercise. Appl Physiol Nutr Metab. 2014 Jul;39(7):787-92. doi: 10.1139/apnm-2013-0507. Epub 2014 Apr 11. PMID 24971679
- [Background] Ortega JF, Hamouti N, Fernandez-Elias VE, de Prada MV, Martinez-Vizcaino V, Mora-Rodriguez R. Metformin does not attenuate the acute insulin-sensitizing effect of a single bout of exercise in individuals with insulin resistance. Acta Diabetol. 2014 Oct;51(5):749-55. doi: 10.1007/s00592-014-0580-4. Epub 2014 Mar 29. PMID 24682492
- [Background] Mora-Rodriguez R, Ortega JF, Hamouti N, Fernandez-Elias VE, Canete Garcia-Prieto J, Guadalupe-Grau A, Saborido A, Martin-Garcia M, Guio de Prada V, Ara I, Martinez-Vizcaino V. Time-course effects of aerobic interval training and detraining in patients with metabolic syndrome. Nutr Metab Cardiovasc Dis. 2014 Jul;24(7):792-8. doi: 10.1016/j.numecd.2014.01.011. Epub 2014 Jan 29. PMID 24656853
- [Background] Diez-Fernandez A, Sanchez-Lopez M, Mora-Rodriguez R, Notario-Pacheco B, Torrijos-Nino C, Martinez-Vizcaino V. Obesity as a mediator of the influence of cardiorespiratory fitness on cardiometabolic risk: a mediation analysis. Diabetes Care. 2014;37(3):855-62. doi: 10.2337/dc13-0416. Epub 2013 Nov 6. PMID 24198304
- [Derived] Alvarez-Jimenez L, Morales-Palomo F, Moreno-Cabanas A, Ortega JF, Mora-Gonzalez D, Mora-Rodriguez R. Acute Statin Withdrawal Does not Interfere With the Improvements of a Session of Exercise in Postprandial Metabolism. J Clin Endocrinol Metab. 2023 Dec 21;109(1):80-91. doi: 10.1210/clinem/dgad477. PMID 37565392
- [Derived] Morales-Palomo F, Moreno-Cabanas A, Alvarez-Jimenez L, Ortega JF, Mora-Rodriguez R. Effect of Yearly Exercise on Medication Expense and Benefit-Cost Ratio in Individuals with Metabolic Syndrome: A Randomized Clinical Trial. Med Sci Sports Exerc. 2023 Feb 1;55(2):158-166. doi: 10.1249/MSS.0000000000003053. Epub 2022 Sep 29. PMID 36171184
- [Derived] Moreno-Cabanas A, Morales-Palomo F, Alvarez-Jimenez L, Ortega JF, Mora-Rodriguez R. Effects of chronic metformin treatment on training adaptations in men and women with hyperglycemia: A prospective study. Obesity (Silver Spring). 2022 Jun;30(6):1219-1230. doi: 10.1002/oby.23410. Epub 2022 May 17. PMID 35578807
- [Derived] Ramirez-Jimenez M, Morales-Palomo F, Moreno-Cabanas A, Alvarez-Jimenez L, Ortega JF, Mora-Rodriguez R. Aerobic exercise training improves nocturnal blood pressure dipping in medicated hypertensive individuals. Blood Press Monit. 2022 Aug 1;27(4):272-275. doi: 10.1097/MBP.0000000000000598. Epub 2022 Apr 18. PMID 35438082
- [Derived] Moreno-Cabanas A, Ortega JF, Morales-Palomo F, Ramirez-Jimenez M, Alvarez-Jimenez L, Mora-Rodriguez R. One Bout of Resistance Training Does Not Enhance Metformin Actions in Prediabetic and Diabetic Individuals. Med Sci Sports Exerc. 2022 Jul 1;54(7):1043-1050. doi: 10.1249/MSS.0000000000002889. Epub 2022 Feb 10. PMID 35142713
- [Derived] Mora-Rodriguez R, Ortega JF, Morales-Palomo F, Ramirez-Jimenez M, Moreno-Cabanas A, Alvarez-Jimenez L. Endurance Exercise Training reduces Blood Pressure according to the Wilder's Principle. Int J Sports Med. 2022 Apr;43(4):336-343. doi: 10.1055/a-1548-6985. Epub 2021 Sep 24. PMID 34560789
- [Derived] Morales-Palomo F, Moreno-Cabanas A, Ramirez-Jimenez M, Alvarez-Jimenez L, Valenzuela PL, Lucia A, Ortega JF, Mora-Rodriguez R. Exercise Reduces Medication for Metabolic Syndrome Management: A 5-Year Follow-up Study. Med Sci Sports Exerc. 2021 Jul 1;53(7):1319-1325. doi: 10.1249/MSS.0000000000002591. PMID 33433153
- [Derived] Alvarez-Jimenez L, Moreno-Cabanas A, Ramirez-Jimenez M, Morales-Palomo F, Ortega JF, Mora-Rodriguez R. Effects of statins and exercise on postprandial lipoproteins in metabolic syndrome vs metabolically healthy individuals. Br J Clin Pharmacol. 2021 Mar;87(3):955-964. doi: 10.1111/bcp.14447. Epub 2020 Jul 12. PMID 32598033
- [Derived] Morales-Palomo F, Ramirez-Jimenez M, Ortega JF, Moreno-Cabanas A, Mora-Rodriguez R. Exercise Training Adaptations in Metabolic Syndrome Individuals on Chronic Statin Treatment. J Clin Endocrinol Metab. 2020 Apr 1;105(4):dgz304. doi: 10.1210/clinem/dgz304. PMID 31875915
- [Derived] Guio de Prada V, Ortega JF, Morales-Palomo F, Ramirez-Jimenez M, Moreno-Cabanas A, Mora-Rodriguez R. Women with metabolic syndrome show similar health benefits from high-intensity interval training than men. PLoS One. 2019 Dec 10;14(12):e0225893. doi: 10.1371/journal.pone.0225893. eCollection 2019. PMID 31821339
- [Derived] Morales-Palomo F, Ramirez-Jimenez M, Ortega JF, Mora-Rodriguez R. Effectiveness of Aerobic Exercise Programs for Health Promotion in Metabolic Syndrome. Med Sci Sports Exerc. 2019 Sep;51(9):1876-1883. doi: 10.1249/MSS.0000000000001983. PMID 31415443
- [Derived] Mora-Rodriguez R, Ortega JF, Ramirez-Jimenez M, Moreno-Cabanas A, Morales-Palomo F. Insulin sensitivity improvement with exercise training is mediated by body weight loss in subjects with metabolic syndrome. Diabetes Metab. 2020 Jun;46(3):210-218. doi: 10.1016/j.diabet.2019.05.004. Epub 2019 May 31. PMID 31158474
- [Derived] Mora-Rodriguez R, Ortega JF, Morales-Palomo F, Ramirez-Jimenez M. Weight loss but not gains in cardiorespiratory fitness after exercise-training predicts improved health risk factors in metabolic syndrome. Nutr Metab Cardiovasc Dis. 2018 Dec;28(12):1267-1274. doi: 10.1016/j.numecd.2018.08.004. Epub 2018 Aug 23. PMID 30459053
- [Derived] Morales-Palomo F, Ramirez-Jimenez M, Ortega JF, Mora-Rodriguez R. Exercise Periodization over the Year Improves Metabolic Syndrome and Medication Use. Med Sci Sports Exerc. 2018 Oct;50(10):1983-1991. doi: 10.1249/MSS.0000000000001659. PMID 29781921
- [Derived] Mora-Rodriguez R, Ramirez-Jimenez M, Fernandez-Elias VE, Guio de Prada MV, Morales-Palomo F, Pallares JG, Nelson RK, Ortega JF. Effects of aerobic interval training on arterial stiffness and microvascular function in patients with metabolic syndrome. J Clin Hypertens (Greenwich). 2018 Jan;20(1):11-18. doi: 10.1111/jch.13130. Epub 2017 Nov 6. PMID 29106772
- [Derived] Mora-Rodriguez R, Fernandez-Elias VE, Morales-Palomo F, Pallares JG, Ramirez-Jimenez M, Ortega JF. Aerobic interval training reduces vascular resistances during submaximal exercise in obese metabolic syndrome individuals. Eur J Appl Physiol. 2017 Oct;117(10):2065-2073. doi: 10.1007/s00421-017-3697-7. Epub 2017 Aug 12. PMID 28803380
- [Derived] Morales-Palomo F, Ramirez-Jimenez M, Ortega JF, Lopez-Galindo PL, Fernandez-Martin J, Mora-Rodriguez R. Effects of repeated yearly exposure to exercise-training on blood pressure and metabolic syndrome evolution. J Hypertens. 2017 Oct;35(10):1992-1999. doi: 10.1097/HJH.0000000000001430. PMID 28594711

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants underwent four trials in a full cross-over randomized fashion. Subject tested before and after 4 months of training. At baseline subjects were tested on two occasions, one with and one without medication separated 72 hours. Post-training testing was similarly conducted with and without medication separated 72 hours.
Groups:
- MEDICATED FIRST THEN PLACEBO: Subjects will remain taking their habitual antihypertensive medication during this time. After this first test, they will receive placebo during 72 h and will be tested again.
- PLACEBO FIRST THEN MEDICATED: Subjects will be withdrawn from their habitual antihypertensive medication during 72 hours, which will be substituted by a placebo. Then their habitual medication will be restated and they will be tested again.
Period: First Intervention Drug Tests
Arm/Group | MEDICATED FIRST THEN PLACEBO | PLACEBO FIRST THEN MEDICATED
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0
Period: Second Intervention Training (4 Months)
Arm/Group | MEDICATED FIRST THEN PLACEBO | PLACEBO FIRST THEN MEDICATED
Started | 20 | 20
Completed | 19 | 19
Not Completed | 1 | 1
Period: Third Intervention Drug Test
Arm/Group | MEDICATED FIRST THEN PLACEBO | PLACEBO FIRST THEN MEDICATED
Started | 19 | 19
Completed | 19 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The baseline trial is the non-medicated, no-exercise
Groups:
- PRE-POST TRAINING: In this cross over design, participants will be tested PRE and POST 4 months of endurance training.
  They will be tested while taking their habitual medication on one occasion and in the other, the investigators will withhold their medication during 72 h to achieve 4 conditions:
  1. Untrained, no medicated.
  2. Untrained, medicated.
  a) Trained, no medicated. b) Trained, medicated.
Arm/Group | PRE-POST TRAINING
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] — Years old rounding up without desmo points BASED ON DATE OF BIRTH
  years | 58.7 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Dichotomic male or female as declared by the own subject
  Participants
    Female | 8
    Male | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — No classification by ethnicity was attempted. In Spain there are more than 25 recognized ethnicities. The program lists Latino or Hispanic as the only choice. However, our subjects do not fit into that category. There are not the product of the mix of races since the discovery and colonization of America starting in 1492 by Spaniards, Portugueses, and Italians. On the contrary, they are the ones that stayed in Europe. The simile will be to stablish that people in US should be named Anglosaxonis.
  Participants
    Hispanic or Latino | 40
    Not Hispanic or Latino | 0
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — In south Europe we have caucasians, asians, blacks, and gypsies as main races. Again, the program does not allow these choices.
  Participants
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 40
    More than one race | 0
    Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants] — The basic region were we are recruiting subjects is south Europe (Spain).
  participants
    Spain | 40

OUTCOME MEASURES:

1. Primary Outcome: Systolic Blood Pressure
Description: Determined using a ECG-gated automated sphygmomanometer. Value is the difference between the placebo and antihypertensive medication.
Time Frame: Subject tested before and after 4 months of training. At baseline tested with and without medication separated 72 hours. Post training tested with and without medication separated 72 hours.
Population: All participants underwent four trials in a full cross-over randomized fashion
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- MEDICATED: Subjects will take their habitual dose of antihypertensive medication.
- PLACEBO: Subjects will be withdrawn from their habitual antihypertensive medication during 72 hours, which will be substituted by a placebo.
Arm/Group | MEDICATED | PLACEBO
Number analyzed (Participants) | 38 | 38
mmHg
  BEFORE TRAINING | 126 (13) | 134 (11)
  AFTER TRAINING | 124 (13) | 133 (12)
Statistical Analysis 1: Comparison: MEDICATED vs PLACEBO; Test type: Other; p = 0.040, ANOVA; repeated measures

2. Primary Outcome: Diastolic Blood Pressure
Description: as for outcome 1
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- MEDICATED: Subjects will be tested while taking their habitual antihypertensive medication.
Arm/Group | MEDICATED | PLACEBO
Number analyzed (Participants) | 38 | 38
mmHg
  BEFORE TRAINING | 75 (8) | 79 (8)
  AFTER TRAINING | 72 (7) | 77 (7)
Statistical Analysis 1: Comparison: MEDICATED vs PLACEBO; Test type: Other; p = 0.054, ANOVA; repeated measures

3. Primary Outcome: Mean Arterial Pressure
Description: as for outcome 1
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | MEDICATED | PLACEBO
Number analyzed (Participants) | 38 | 38
mmHg
  BEFORE TRAINING | 92 (9) | 97 (8)
  AFTER TRAINING | 89 (8) | 96 (8)
Statistical Analysis 1: Comparison: MEDICATED vs PLACEBO; Test type: Other; p = 0.040, ANOVA; REPEATED MEASURES

4. Secondary Outcome: Maximal Oxygen Consumption Rate During Exercise (VO2max).
Description: Index of cardiorespiratory fitness assessed during an incremental cycle-ergometer test using an indirect calorimetry system.
  Value is the difference between the placebo and antihypertensive medication.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters of O2/kg weight/min
Arm/Group | MEDICATED | PLACEBO
Number analyzed (Participants) | 38 | 38
Liters of O2/kg weight/min
  BEFORE TRAINING | 2.26 (0.58) | 2.26 (0.58)
  AFTER TRAINING | 2.49 (0.55) | 2.49 (0.55)
Statistical Analysis 1: Comparison: MEDICATED vs PLACEBO; Test type: Other; p = 0.321, ANOVA; REPEATED MEASURES

5. Secondary Outcome: Maximal Rate of Fat Oxidation.
Description: Calculated in grams per min during the incremental cycloergometer test wih the use of indirect calorimetry system.
  Value is the difference between the placebo and antihypertensive medication.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: grams/min
Arm/Group | MEDICATED | PLACEBO
Number analyzed (Participants) | 38 | 38
grams/min
  BEFORE TRAINING | 0.24 (0.10) | 0.24 (0.10)
  AFTER TRAINING | 0.28 (0.15) | 0.28 (0.15)
Statistical Analysis 1: Comparison: MEDICATED; Test type: Other; p = 0.401, ANOVA; REPEATED MEASURES

6. Secondary Outcome: Body Weight
Description: Nude body weight. Value is the difference between the placebo and antihypertensive medication.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | MEDICATED | PLACEBO
Number analyzed (Participants) | 38 | 38
kg
  BEFORE TRAINING | 92.1 (13.6) | 92.5 (13.6)
  AFTER TRAINING | 90.0 (13.2) | 90.8 (13.4)
Statistical Analysis 1: Comparison: MEDICATED; Test type: Other; p = 0.021, ANOVA; REPEATED MEASURES

ADVERSE EVENTS:
Time Frame: 4 months of the intervention
Description: No adverse events were recorded
Groups:
- MEDICATED vs NO MEDICATED BEFORE TRAINING: Subjects will be tested twice one taking their habitual dose of medication, and in the other, the investigators will withhold their medication during 72 h.
  1. Untrained, no medicated.
  2. Untrained, medicated.
- MEDICATED vs NO MEDICATED AFTER EXERCISE TRAINING: After 4 months of endurance training subjects will be tested twice one taking their habitual dose of medication, and in the other, the investigators will withhold their medication during 72 h.
  c) Trained, no medicated. d) Trained, medicated.
Arm/Group | MEDICATED vs NO MEDICATED BEFORE TRAINING | MEDICATED vs NO MEDICATED AFTER EXERCISE TRAINING
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2017-08-30): https://cdn.clinicaltrials.gov/large-docs/96/NCT03019796/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-30): https://cdn.clinicaltrials.gov/large-docs/96/NCT03019796/SAP_001.pdf
  • Informed Consent Form (2017-08-30): https://cdn.clinicaltrials.gov/large-docs/96/NCT03019796/ICF_002.pdf